CLINICAL TRIAL: NCT03778658
Title: AYA-UNITE (Utilizing Novel Information Technology to Promote Exercise and Well-Being)
Brief Title: Utilizing Novel Information Technology to Promote Exercise and Well-Being in Adolescents and Young Adults With Cancer
Acronym: AYA-UNITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Pooja Rao, Pooja Rao, M.D. , Assistant Professor, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00010118
Record Dates: First submitted 2018-12-13; First posted 2018-12-19 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Adolescent; Young Adult; Cancer; Physical Activity; Psychological Distress; Social Isolation
Keywords: Adolescent/Young Adult; Cancer; Physical Activity; Psychosocial Health
MeSH Terms: conditions — Neoplasms; Motor Activity; Social Isolation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Outpatient Physical Activity Program (Experimental): The intervention will investigate a multi modal outpatient physical activity program incorporating both strength training utilizing resistance bands, as well as an aerobic activity based on hip-hop dancing.
  Interventions: Behavioral: Physical Activity Intervention

INTERVENTIONS:
Behavioral: Physical Activity Intervention — Participants will engage in a multimodal aerobic and strength training intervention.

SUMMARY:
Adolescents and young adults (AYAs) with cancer have many needs for supportive care that differ from younger and older patients.This includes age-appropriate psychological support for management of distress, as well as supports for the social isolation many AYAs experience. One intervention that may provide AYAs with cancer improved psychosocial support, as well as increased physical strength, is physical activity. This feasibility project aims to evaluate the safety, feasibility and acceptability of a physical activity training in AYAs with cancer delivered via a socially interactive videoconferencing platform.

DETAILED DESCRIPTION:
Adolescents and young adults (AYAs) with cancer comprise a unique population within the larger cancer community. This is primarily due to distinct differences in disease biology compared to older and younger patients, as well as their unique psychosocial needs. AYAs with cancer historically have unmet needs relating to management of their mental health and treatment-related symptoms. One particular area of unmet need is distress management during cancer treatment, reported in nearly one third of AYAs with newly diagnosed cancer. Reasons for distress are multifactorial, including lack of medical information, worries about future life goals and fertility, and social isolation from peers and family. Proactively addressing and preventing this distress is critical for forestalling the high rates of depression, anxiety, and post-traumatic stress seen in AYAs. One promising but under explored intervention with the potential to mitigate distress is group-based physical activity. Multiple studies cite physical activity's benefits for patients with cancer, while oncology and sports medicine societies recommend including physical activity as part of comprehensive cancer care. Group physical activity intervention models have been successful in creating sustainable improvements in physical and psychosocial health in other populations with cancer, though can present transportation and scheduling barriers. Additionally, medical providers and participants undergoing treatment for cancer may be hesitant to engage in group-based physical activity interventions during times of neutropenia given infection risk.

Dr. Rao's mentors have extensive preliminary data that guided her project's development. The theoretical model for this study's intervention delivery is based on Dr. Rovniak's Social Networks for Activity Promotion (SNAP) model, and targets optimizing the physical environment where physical activity is received, as well as the importance of social network environments and interactions. Dr. Schmitz has been at the forefront of the movement to incorporate physical activity into the care of patients with cancer and cancer survivors. She has led multiple trials, including a large randomized controlled trial to assess the safety of upper body exercise among breast cancer survivors with and without lymphedema (Physical Activity and Lymphedema Trial [PAL]). Dr. Sciamanna's work has evaluated the implementation of a group strength training intervention in elderly patients, which has been found to be safe and effective, as well socially beneficial to its participants. Dr. Williams is the founder and president of Hip Hop for Public Health (HHPH) a non-profit organization which has successfully utilized hip-hop music to deliver sustainable health messages pertaining to nutrition and physical activity in youth.

The preliminary data as noted above set the foundation for this project, which builds on the importance of social network environments and interactions in encouraging physical activity. This is particularly true for adolescents as a whole, as social support has been found to be an especially important factor in the promotion of physical activity. Specifically for AYAs with cancer, physical activity has been cited as an area of preferred clinical program focus for AYAs with cancer and those who have completed treatment. Thus, a group-based physical activity intervention among AYAs with cancer could address an area of unmet need that potentially improves the psychosocial health of this patient population. Delivery using a virtual platform is culturally appropriate for AYAs with cancer, a unique patient population that is technologically savvy, and interested in using social media platforms to create a sense of belonging and community.

ELIGIBILITY:
Inclusion Criteria:

* Participant age 15-21 years old at time of cancer diagnosis
* Participant diagnosis of cancer who is currently undergoing active treatment for cancer, or who is within 3 years of end of cancer treatment at the time of enrollment
* Participant receiving oncologic care at Penn State Health Children's Hospital or Penn State Cancer Institute
* Participant fluency in written and spoken English for participants >= 18 years old
* Parent and participant fluency in written and spoken English for participants < 18 years old
* Primary attending oncologist approval
* Participant must have access to a computer or smartphone
* Performance status of ECOG <= 2, and Lansky /Karnofsky scale >= 50

Exclusion Criteria:

* Cardiovascular or respiratory disease
* Class II, III or IV heart failure as defined by the New York Heart Association functional classification system
* History of acute coronary syndromes (including myocardial infarction and unstable angina), coronary angioplasty or stenting within the past 6 months prior to the start of chemotherapy
* Uncontrolled arrhythmias
* Syncope
* Acute myocarditis, pericarditis or endocarditis
* Diagnosed with pulmonary embolism or pulmonary infarction within 3 months of enrollment
* Diagnosed with deep venous thrombosis within 3 months of enrollment
* Any history of intracardiac thrombosis
* Suspected dissecting aneurysm
* Pulmonary edema
* Respiratory failure
* Acute non-cardiopulmonary disorder that may affect exercise performance or be exacerbated by physical activity
* Altered mental status or dementia
* Mental impairment leading to inability to cooperate
* Active bleeding
* Absolute contraindication to exercise
* Hemodynamic instability
* Pregnant women
* Non-English speaking
* Recent initiation of physical activity program within last 3 months
* Patients with relapsed cancer
* Patients who have undergone allogeneic stem cell transplant

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Safety | Weekly during 12 week study
  Proportion of participants experiencing musculoskeletal (MSK) impairment, adverse effects requiring treatment alterations, and injury rate for MSK injuries (defined as symptoms lasting 1 week or longer and/or requiring attention of provider)
Feasibility | At end of 12 week study
  Physical activity intervention arm will be considered feasible if at least 50% of the participants complete 80% of the training sessions.
Acceptability | At end of 12 week study
  The physical activity intervention will be considered acceptable if more than 50% of the approached participants agree to receive at least the first session of the physical activity intervention.

SECONDARY OUTCOMES:
Physical function assessments: Arm curl test of dominant arm (tests upper body strength) | Baseline and at end of 12 week study
  Arm curl test assessment will be performed on all participants using free weights of 5 lb and 8 lb (or household alternative object)
Physical function assessments: 30-second Chair Stand (tests leg strength and endurance) | Baseline and at end of 12 week study
  The 30-second Chair Stand will be performed on all participants
Physical function assessments: Timed Up and Go (tests mobility) | Baseline and at end of 12 week study
  The Timed Up and Go test will be performed on all participants
Physical function assessments: 4-Stage Balance (tests balance) | Baseline and at end of 12 week study
  The 4-Stage Balance will be performed on all participants
Physical function assessments: Patient reported physical function | Baseline and at end of 12 week study
  Physical function: The Patient-Reported Outcomes Measurement Information System (PROMIS)
Psychosocial measurements: Distress | Baseline and at end of 12 week study
  Distress: The Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Psychological Stress Experiences Form will be used.
Psychosocial measurements: Social Isolation | Baseline and at end of 12 week study
  Social Isolation: The Patient-Reported Outcomes Measurement Information System (PROMIS) Item Bank Social Isolation Short Form 8a will be used.
Psychosocial measurements: Fatigue | Baseline and at end of 12 week study
  Fatigue: The Patient-Reported Outcomes Measurement Information System (PROMIS) Cancer Item Bank v1.0- Fatigue will be used.
Psychosocial measurements: Quality of Life | Baseline and at end of 12 week study
  Quality of Life: The Patient-Reported Outcomes Measurement Information System (PROMIS) PROMIS-29 Profile will be used.
Patient-reported symptoms | All participants will be given this instrument once prior to study initiation, and once every 3 weeks during the study.
  PRO-CTCAE will be used to collect and measure information of patient-PRO-CTCAE will be used to collect and measure information of patient-reported symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Rao, MD MSCE, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmitz KH, Ahmed RL, Troxel A, Cheville A, Smith R, Lewis-Grant L, Bryan CJ, Williams-Smith CT, Greene QP. Weight lifting in women with breast-cancer-related lymphedema. N Engl J Med. 2009 Aug 13;361(7):664-73. doi: 10.1056/NEJMoa0810118. PMID 19675330
- [Background] Powell KE, Heath GW, Kresnow MJ, Sacks JJ, Branche CM. Injury rates from walking, gardening, weightlifting, outdoor bicycling, and aerobics. Med Sci Sports Exerc. 1998 Aug;30(8):1246-9. doi: 10.1097/00005768-199808000-00010. PMID 9710864
- [Background] Courneya KS, McKenzie DC, Reid RD, Mackey JR, Gelmon K, Friedenreich CM, Ladha AB, Proulx C, Lane K, Vallance JK, Segal RJ. Barriers to supervised exercise training in a randomized controlled trial of breast cancer patients receiving chemotherapy. Ann Behav Med. 2008 Feb;35(1):116-22. doi: 10.1007/s12160-007-9009-4. Epub 2008 Feb 20. PMID 18347912
- [Background] Zhang X, McClean D, Ko E, Morgan MA, Schmitz K. Exercise Among Women With Ovarian Cancer: A Feasibility and Pre-/Post-Test Exploratory Pilot Study. Oncol Nurs Forum. 2017 May 1;44(3):366-374. doi: 10.1188/17.ONF.366-374. PMID 28635971
- [Background] Hinds PS, Nuss SL, Ruccione KS, Withycombe JS, Jacobs S, DeLuca H, Faulkner C, Liu Y, Cheng YI, Gross HE, Wang J, DeWalt DA. PROMIS pediatric measures in pediatric oncology: valid and clinically feasible indicators of patient-reported outcomes. Pediatr Blood Cancer. 2013 Mar;60(3):402-8. doi: 10.1002/pbc.24233. Epub 2012 Jul 24. PMID 22829446
- [Background] Henderson JR 2nd, Kiernan E, McNeer JL, Rodday AM, Spencer K, Henderson TO, Parsons SK. Patient-Reported Health-Related Quality-of-Life Assessment at the Point-of-Care with Adolescents and Young Adults with Cancer. J Adolesc Young Adult Oncol. 2018 Feb;7(1):97-102. doi: 10.1089/jayao.2017.0046. Epub 2017 Nov 30. PMID 29190179
- [Background] Warner EL, Kent EE, Trevino KM, Parsons HM, Zebrack BJ, Kirchhoff AC. Social well-being among adolescents and young adults with cancer: A systematic review. Cancer. 2016 Apr 1;122(7):1029-37. doi: 10.1002/cncr.29866. Epub 2016 Feb 5. PMID 26848713
- [Background] Barakat LP, Galtieri LR, Szalda D, Schwartz LA. Assessing the psychosocial needs and program preferences of adolescents and young adults with cancer. Support Care Cancer. 2016 Feb;24(2):823-832. doi: 10.1007/s00520-015-2849-8. Epub 2015 Jul 21. PMID 26190361
- [Background] Muffly LS, Hlubocky FJ, Khan N, Wroblewski K, Breitenbach K, Gomez J, McNeer JL, Stock W, Daugherty CK. Psychological morbidities in adolescent and young adult blood cancer patients during curative-intent therapy and early survivorship. Cancer. 2016 Mar 15;122(6):954-61. doi: 10.1002/cncr.29868. Epub 2016 Jan 7. PMID 26749023
- [Background] Quinn GP, Goncalves V, Sehovic I, Bowman ML, Reed DR. Quality of life in adolescent and young adult cancer patients: a systematic review of the literature. Patient Relat Outcome Meas. 2015 Feb 17;6:19-51. doi: 10.2147/PROM.S51658. eCollection 2015. PMID 25733941
- [Background] Burgoyne MJ, Bingen K, Leuck J, Dasgupta M, Ryan P, Hoffmann RG. Cancer-Related Distress in Young Adults Compared to Middle-Aged and Senior Adults. J Adolesc Young Adult Oncol. 2015 Jun;4(2):56-63. doi: 10.1089/jayao.2014.0005. Epub 2015 Jun 2. PMID 26812552
- [Background] McCarthy MC, McNeil R, Drew S, Orme L, Sawyer SM. Information needs of adolescent and young adult cancer patients and their parent-carers. Support Care Cancer. 2018 May;26(5):1655-1664. doi: 10.1007/s00520-017-3984-1. Epub 2017 Dec 8. PMID 29222598
- [Background] McCarthy MC, McNeil R, Drew S, Dunt D, Kosola S, Orme L, Sawyer SM. Psychological Distress and Posttraumatic Stress Symptoms in Adolescents and Young Adults with Cancer and Their Parents. J Adolesc Young Adult Oncol. 2016 Dec;5(4):322-329. doi: 10.1089/jayao.2016.0015. Epub 2016 May 23. PMID 27214245
- [Background] Kwak M, Zebrack BJ, Meeske KA, Embry L, Aguilar C, Block R, Hayes-Lattin B, Li Y, Butler M, Cole S. Trajectories of psychological distress in adolescent and young adult patients with cancer: a 1-year longitudinal study. J Clin Oncol. 2013 Jun 10;31(17):2160-6. doi: 10.1200/JCO.2012.45.9222. Epub 2013 May 6. PMID 23650425
- [Background] Kwak M, Zebrack BJ, Meeske KA, Embry L, Aguilar C, Block R, Hayes-Lattin B, Li Y, Butler M, Cole S. Prevalence and predictors of post-traumatic stress symptoms in adolescent and young adult cancer survivors: a 1-year follow-up study. Psychooncology. 2013 Aug;22(8):1798-806. doi: 10.1002/pon.3217. Epub 2012 Nov 8. PMID 23135830
- [Background] Cormie P, Zopf EM, Zhang X, Schmitz KH. The Impact of Exercise on Cancer Mortality, Recurrence, and Treatment-Related Adverse Effects. Epidemiol Rev. 2017 Jan 1;39(1):71-92. doi: 10.1093/epirev/mxx007. PMID 28453622
- [Background] Schmitz KH, Courneya KS, Matthews C, Demark-Wahnefried W, Galvao DA, Pinto BM, Irwin ML, Wolin KY, Segal RJ, Lucia A, Schneider CM, von Gruenigen VE, Schwartz AL; American College of Sports Medicine. American College of Sports Medicine roundtable on exercise guidelines for cancer survivors. Med Sci Sports Exerc. 2010 Jul;42(7):1409-26. doi: 10.1249/MSS.0b013e3181e0c112. PMID 20559064
- [Background] Wolin KY, Schwartz AL, Matthews CE, Courneya KS, Schmitz KH. Implementing the exercise guidelines for cancer survivors. J Support Oncol. 2012 Sep-Oct;10(5):171-7. doi: 10.1016/j.suponc.2012.02.001. Epub 2012 May 10. PMID 22579268
- [Background] Rovniak LS, Sallis JF, Kraschnewski JL, Sciamanna CN, Kiser EJ, Ray CA, Chinchilli VM, Ding D, Matthews SA, Bopp M, George DR, Hovell MF. Engineering online and in-person social networks to sustain physical activity: application of a conceptual model. BMC Public Health. 2013 Aug 14;13:753. doi: 10.1186/1471-2458-13-753. PMID 23945138
- [Background] Rovniak LS, Kong L, Hovell MF, Ding D, Sallis JF, Ray CA, Kraschnewski JL, Matthews SA, Kiser E, Chinchilli VM, George DR, Sciamanna CN. Engineering Online and In-Person Social Networks for Physical Activity: A Randomized Trial. Ann Behav Med. 2016 Dec;50(6):885-897. doi: 10.1007/s12160-016-9814-8. PMID 27405724
- [Background] Sciamanna CN, Patel VA, Kraschnewski JL, Rovniak LS, Messina DA, Stuckey HL, Curry WJ, Chuang CH, Sherwood LL, Hess SL. A strength training program for primary care patients, central Pennsylvania, 2012. Prev Chronic Dis. 2014 Jun 26;11:E107. doi: 10.5888/pcd11.130403. PMID 24967829
- [Background] Schmitz KH, Troxel AB, Cheville A, Grant LL, Bryan CJ, Gross CR, Lytle LA, Ahmed RL. Physical Activity and Lymphedema (the PAL trial): assessing the safety of progressive strength training in breast cancer survivors. Contemp Clin Trials. 2009 May;30(3):233-45. doi: 10.1016/j.cct.2009.01.001. Epub 2009 Jan 8. PMID 19171204
- [Background] Schmitz KH, Ahmed RL, Troxel AB, Cheville A, Lewis-Grant L, Smith R, Bryan CJ, Williams-Smith CT, Chittams J. Weight lifting for women at risk for breast cancer-related lymphedema: a randomized trial. JAMA. 2010 Dec 22;304(24):2699-705. doi: 10.1001/jama.2010.1837. Epub 2010 Dec 8. PMID 21148134
- [Background] Williams O, Leighton-Herrmann E, DeSorbo A, Hecht M, Hedmann M, Huq S, Gerin W, Chinchilli V, Ogedegbe G, Noble J. Hip Hop Stroke: Study Protocol for a Randomized Controlled Trial to Address Stroke Literacy. J Clin Trials. 2015 Oct;5(5):242. doi: 10.4172/2167-0870.1000242. Epub 2015 Oct 23. PMID 26779395
- [Background] Williams O, Leighton-Herrmann Quinn E, Teresi J, Eimicke JP, Kong J, Ogedegbe G, Noble J. Improving Community Stroke Preparedness in the HHS (Hip-Hop Stroke) Randomized Clinical Trial. Stroke. 2018 Apr;49(4):972-979. doi: 10.1161/STROKEAHA.117.019861. PMID 29567762
- [Background] Mendonca G, Cheng LA, Melo EN, de Farias Junior JC. Physical activity and social support in adolescents: a systematic review. Health Educ Res. 2014 Oct;29(5):822-39. doi: 10.1093/her/cyu017. Epub 2014 May 8. PMID 24812148
- [Background] Cheung CK, Zebrack B. What do adolescents and young adults want from cancer resources? Insights from a Delphi panel of AYA patients. Support Care Cancer. 2017 Jan;25(1):119-126. doi: 10.1007/s00520-016-3396-7. Epub 2016 Aug 31. PMID 27580714
- [Background] Perales MA, Drake EK, Pemmaraju N, Wood WA. Social Media and the Adolescent and Young Adult (AYA) Patient with Cancer. Curr Hematol Malig Rep. 2016 Dec;11(6):449-455. doi: 10.1007/s11899-016-0313-6. PMID 26893061
- [Background] Schmitz KH. Incorporating Strength Training into Cancer Care: Translating PAL into the Strength After Breast Cancer Program. Obesity (Silver Spring). 2017 Nov;25 Suppl 2:S32-S33. doi: 10.1002/oby.22018. No abstract available. PMID 29086524
- [Background] Ness KK, Baker KS, Dengel DR, Youngren N, Sibley S, Mertens AC, Gurney JG. Body composition, muscle strength deficits and mobility limitations in adult survivors of childhood acute lymphoblastic leukemia. Pediatr Blood Cancer. 2007 Dec;49(7):975-81. doi: 10.1002/pbc.21091. PMID 17091482
- [Background] Teodozio CGC, Chaves GV, Arcuri IP, Frajacomo FT. Does grip strength decrease in the very early stages of hematological treatment? Support Care Cancer. 2018 Feb;26(2):333-335. doi: 10.1007/s00520-017-3932-0. Epub 2017 Oct 23. PMID 29058129
- [Background] Bourdon A, Grandy SA, Keats MR. Aerobic exercise and cardiopulmonary fitness in childhood cancer survivors treated with a cardiotoxic agent: a meta-analysis. Support Care Cancer. 2018 Jul;26(7):2113-2123. doi: 10.1007/s00520-018-4208-z. Epub 2018 Apr 18. PMID 29671063
- [Background] Reeve BB, McFatrich M, Pinheiro LC, Freyer DR, Basch EM, Baker JN, Withycombe JS, Sung L, Mack JW, Waldron MK, Mowbray C, Palma D, Hinds PS. Cognitive Interview-Based Validation of the Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events in Adolescents with Cancer. J Pain Symptom Manage. 2017 Apr;53(4):759-766. doi: 10.1016/j.jpainsymman.2016.11.006. Epub 2017 Jan 3. PMID 28062347
- [Derived] Rao P, Kazak AE, Doerksen SE, Koehly LM, Verdery AM, Heitzenrater J, Harding BA, Byrnes CL, Costigan HJ, Rovniak LS, Sciamanna CN, Van Scoy LJ, Schmitz KH. AYA-UNITE: Lessons Learned on Intervention Development Promoting Social and Physical Health of Adolescent/Young Adult Cancer Survivors. J Adolesc Young Adult Oncol. 2023 Dec;12(6):929-934. doi: 10.1089/jayao.2023.0093. Epub 2023 Oct 9. PMID 37815633